CLINICAL TRIAL: NCT07088055
Title: Multi-center, 6-month, Randomized, and Controlled Trial to Compare the Effects of Myo Munchee Therapy and Oral Motor Therapy (OMT) in Pediatric Patients (Aged 3-5 Years) to Treat Maxillary Deficiency and Orofacial Myofunctional Dysfunction (OMD).
Brief Title: Trial to Compare the Effects of Myo Munchee Therapy and Oral Motor Therapy (OMT) in Pediatric Patients to Treat Maxillary Deficiency and Orofacial Myofunctional Dysfunction (OMD).
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Myo Munchee (Operations) Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0001
Record Dates: First submitted 2025-06-26; First posted 2025-07-28 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Orofacial Myofunctional Disorders; Myo Munchee; Oral Motor Therapy; Maxillary Deficiency
MeSH Terms: conditions — Retrognathia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (4):
- Control group (No Intervention): There will be no intervention administered to this group. This group will have their clinical and questionnaire measurements taken at the beginning, week 10 and week 26 of the study.
- Myo Munchee Only (Experimental): This group will be administered the Myo Munchee and be given a protocol to follow over the 26-week study period. They will also have the clinical and questionnaire measurements taken at the beginning, week 10 and week 26 of the study.
  Interventions: Device: Chewing device only
- Oral Motor Therapy Only (Active Comparator): This group will be administered an Oral Motor Therapy program to follow over the 26-week study period. They will also have the clinical and questionnaire measurements taken at the beginning, week 10 and week 26 of the study.
  Interventions: Other: Oral Motor Therapy Treatment Arm
- Myo Munchee and Oral Motor Therapy (Active Comparator): This group will be administered an Oral Motoro Therapy program as well as a Myo Munchee protocol to follow over the 26-week study period. They will also have the clinical and questionnaire measurements taken at the beginning, week 10 and week 26 of the study.
  Interventions: Device: Myo Munchee and Oral Motor Therapy Treatment

INTERVENTIONS:
Device: Chewing device only — This group will be administered the Myo Munchee and be given a protocol to follow over the 26-week study period. They will also have the clinical and questionnaire measurements taken at the beginning, week 10 and week 26 of the study.
  Other Names: Chewing device
  Arms: Myo Munchee Only
Device: Myo Munchee and Oral Motor Therapy Treatment — This group will be administered an Oral Motoro Therapy program as well as a Myo Munchee protocol to follow over the 26-week study period. They will also have the clinical and questionnaire measurements taken at the beginning, week 10 and week 26 of the study.
  Other Names: Chewing device; Oral Motor Therapy
  Arms: Myo Munchee and Oral Motor Therapy
Other: Oral Motor Therapy Treatment Arm — This group will be administered an Oral Motor Therapy program to follow over the 26-week study period. They will also have the clinical and questionnaire measurements taken at the beginning, week 10 and week 26 of the study.
  Other Names: Oral Motor Therapy
  Arms: Oral Motor Therapy Only

SUMMARY:
Multi-center, 6-month, randomized, and controlled trial to compare the effects of Myo Munchee therapy and Oral Motor Therapy (OMT) in pediatric patients (aged 3-5 years) to treat maxillary deficiency and orofacial myofunctional dysfunction (OMD).

DETAILED DESCRIPTION:
This study is intended for 3-5 year old children who have a deficiency in their maxillary, dental and oral muscle development. They are at the ideal age for undertaking preventative dental and Oral Motor Therapy to improve their orofacial (referring to structures in the mouth, jaw, lips and cheeks) development, which will likely improve their health and wellbeing. The therapies being used are Oral Motor Therapy and Myo Munchee Therapy. Oral Motor Therapy is a type of therapy used by Speech-Language Pathologists to help patients with feeding, chewing and swallowing difficulties. The Myo Munchee, is a small handheld medical device that fits within the mouth. It is intended for children that have issues with (a) dribbling and drooling, mouth breathing in the daytime or during sleep, (c) messy eating, (d) misaligned teeth, (e) ear and sinus congestion, and (f) teeth clenching and grinding. Both of these therapies are clinically effective and safe. They are low-cost and minimally invasive treatments to resolve OMD's (referring to abnormal patterns of movement, function or positioning of the muscles of the mouth, face, and jaw that interfere with normal growth, development or function) and likely improve maxillary deficiency (referring to the underdevelopment or abnormality of the upper jaw).

ELIGIBILITY:
Inclusion Criteria:

* Aged between 36 - 60 (3-5 yrs) months old and will not turn 6 years of age before the study completion
* Diagnosed with having at least two maxillary skeletal-dental malocclusion traits as determined by the dentist
* At least one of the identified Orofacial Myofunctional Dysfunction (OMD) traits determined by the Speech-Language Pathologist (CCC-SLP)

Exclusion Criteria:

* A patient must be considered healthy to be included in this study. Definition of health: the patient does not have ongoing treatment, medication or specialized assessments (more than routine follow up exams) with health care providers regarding a condition. If they have had treatment for a condition (e.g. treated by respiratory physician for acute asthma hospitalization), it must have been 12 months or more since their last appointment with a health provider related to that condition.

Of particular consideration:

Ongoing care from a sleep physician or respiratory physician Current use of Continuous Positive Airway Pressure (CPAP), nasal sprays, sleeping or behavioral medication to treat diagnosed sleep disorder or behavioral disorder Adenectomy or tonsillectomy within last 12 months

* Any previous or current tumors or traumas in the head, neck and jaw region Patients with any known genetic or congenital conditions that impair oral motor muscle function, oral motor coordination, or speech articulation, such as but not limited to muscular dystrophy, cerebral palsy, will be excluded from the study.
* Patients with any known syndromic conditions to affect oral motor function, including but not limited to syndromes that involve craniofacial anomalies, neuromuscular disorders, or developmental delays affecting oral motor muscle control, speech articulation, or swallowing, such as Down Syndrome, Pierre Robin sequence, or Moebius syndrome.
* Children that do not have their 2nd molars by 36 months of age
* Overweight, Z-scores Body Mass Index (BMI) above 85th percentile (z score of 1) Boys: https://www.cdc.gov/growthcharts/data/extended-bmi/BMI-Age-percentiles-BOYS-Z-Scores.pdf Girls: https://www.cdc.gov/growthcharts/data/extended-bmi/BMI-Age-percentiles-GIRLS-Z-Scores.pdf
* History of prescription for therapeutic gum chewing and/or use of edibles in treatment program
* Previous tongue tie releases (frenuloplasty and frenectomy)
* Any therapeutic oral device treatment
* Previous or current treatment from any other dental, Oral Motor Therapy (OMT) or orthodontic provider
* Gross neglect of patient's oral health and presence of dental caries
* Grade 4 tonsils on Brodsky scale

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 48 (Estimated)
Dates: Start 2025-08-20 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Maxillary expansion | 26 weeks
  1. Palatal transverse width (in mm) expansion. Measured using an intraoral 3D iTero scanner.
  2. Palatal sagittal depth (in mm) expansion. Measured using an intraoral 3D iTero scanner.
  3. Palatal vault height (in mm) expansion. Intraoral measurements taken using an intraoral 3D iTero scanner, which is used to print a 3D model of the intraoral maxilla. The palatal height will then be measured using a GPM & Holtain Palatometer (Model no. 215)

SECONDARY OUTCOMES:
Resolution of dysfunctional resting mouth posture | 26 weeks
  Resting mouth posture outcome will be considered resolved if the below measurements are no longer present at the final evaluation. To assess this outcome, the Speech-Language Pathologist (SLP) will assess if:
  1. Lips open when the child is resting
  2. Mouth breathing during the day and night as mentioned by parent
  3. Tongue rests on the floor of the mouth. The SLP will gently pull down the chin at rest and again look to see where the tongue is once the lips have opened. This is performed after movement, eating and while the patient is sitting.
  If any of these parameters is present at the first evaluation and then resolved at the final evaluation (i.e. no longer present), this will be consider a completed secondary outcome.
Resolution of Oral Motor Development Sequence dysfunction | 26 weeks
  Oral Motor Development Sequence dysfunction will be determined by the SLP against 6 parameters, which is expected of a child to be able to do by 36 months of age:
  1. Internal jaw stabilization
  2. Tongue-tip elevation for swallowing
  3. Appropriate jaw grading for biting and chewing
  4. Gradual refinement of tongue movements
  5. Circular rotary chew patterns
  6. Mature swallow pattern
  The above criteria will be measured during the initial evaluation and determined if they have dysfunction in any of the domains (1-6). They will then be reassessed at 26 weeks during the final evaluation and assess if they have been resolved after completing the study's intervention.
Improvement in patients sleep and behavior | 26 weeks
  Improvement in sleep and behavior as evaluated with the Children's General Airway Screening Protocol (C-GASP) Questionnaire.
Improvement in patients sleep and behavior | 26 weeks
  Improvement in sleep and behavior as evaluated with the Sleep Disorders Inventory for Students-Revised (SDIS-R) by Child Uplift, Inc

CONTACTS AND LOCATIONS:
Overall Officials: Ignatius Bourke, Bachelor of Science (Hons), Principal Investigator — Myo Munchee (Operations) Pty Ltd
Locations (2):
- United States (2):
  - Center for Svedhyaya Therapy Services, Chicago, Illinois
  - Dentistry for Children, Chicago, Illinois

IPD SHARING:
Plan to Share IPD: No
The individual participant data will only be shared with those researchers involved in the study. Specifically, the clinicians who will be taking the measurements and administering the therapy will have access to the de-identified data. The Principal Investigator will also have access to the de-identified data. No other person or persons will have access to the de-identified data.

REFERENCES:
- [Background] Thilander B. Dentoalveolar development in subjects with normal occlusion. A longitudinal study between the ages of 5 and 31 years. Eur J Orthod. 2009 Apr;31(2):109-20. doi: 10.1093/ejo/cjn124. PMID 19304760
- See also: Myo Munchee Homepage — https://myomunchee.com/
- See also: Myo Munchee Educational Material — https://drive.google.com/drive/folders/1gI8FREl1xU1-2jF6NQLFtHGfgMYGnyZ1
- See also: Oral Motor Therapy Exercises — https://www.youtube.com/watch?v=E1tG8ievCig&list=PL-123PNzwf0kaNOfTFzExubUx4XssAXfo

DOCUMENTS (1):
  • Study Protocol (2025-04-25): https://cdn.clinicaltrials.gov/large-docs/55/NCT07088055/Prot_000.pdf